CLINICAL TRIAL: NCT05002660
Title: Evaluation of a Civic Engagement Approach to Catalyze Built Environment Change and Promote Healthy Eating and Physical Activity Among Rural Residents
Brief Title: The Change Club Study: Evaluation of Civic Engagement for Built Environment Change and Health Improvement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Cornell University (Other); Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA230738 (NIH)
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Heart Diseases
Keywords: Physical Activity; Built Environment; Eating Habits
MeSH Terms: conditions — Heart Diseases; Motor Activity; Feeding Behavior | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Community-based cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Intervention) (Experimental): For Change Club members (CCM) only: CCM will participate in meetings of the Change Club and continue implementation of a change to the community environment for up to an additional 24 months. Change Club members will also be asked to recruit 10 or more friends and family members (FFM) to participate in the research study.
  In addition, 100 community residents (CR) will be recruited into the study. Family members, friends and community residents do not participate in the Change Club, but may hear about Change Club activities in their community.
  Interventions: Behavioral: Group 1 (Intervention)
- Group 2 (Control) (Experimental): Control group participants will participate in no intervention activities during the 3-year research study.
  Interventions: Behavioral: Group 2 (Control)

INTERVENTIONS:
Behavioral: Group 1 (Intervention) — The investigators will evaluate the efficacy of the CC curriculum in a 24-months community-based randomized controlled trial. They will compare changes in CVD-related anthropometric, behavioral, and psychosocial parameters between subjects in intervention and control communities.
  Arms: Group 1 (Intervention)
Behavioral: Group 2 (Control) — Group 2 will be offered the same activities as Group 1 after the conclusion of the research study.
  Arms: Group 2 (Control)

SUMMARY:
This is a community randomized controlled trial to evaluate a civic engagement curriculum through which residents will identify barriers and facilitators to healthy eating and physical activity and then implement a project in their communities.

DETAILED DESCRIPTION:
The purpose of this research is to better understand how resident-led activities to change the community environment affect health. The Change Club is a small group of residents who will try to change their community environment relative to food (for example, foods in restaurants or schools) or physical activity opportunities (for example, parks or walking trails) by following a step-wise process facilitated by an extension educator. The purpose of this research is to better understand if and how these activities affect individual behaviors (for example physical activity) and health outcomes (for example BMI) of adults in rural communities.

This study will take place in designated rural communities in Texas and New York. It is planned that about 2,260 people will participate in this study. Some will participate as Change Club members; some will participate as family and friends of Change Club members; and others will participate as community residents.

ELIGIBILITY:
Inclusion Criteria:

We will be recruiting Change Club members (CCM), friend and family members (FFM) of CCM, and community residents (CR).

Common inclusion criteria include:

* Age 18-99
* English-speaking

CCM also must:

* Provide consent electronically
* Be willing to be randomized to either group
* Score "poor" or "intermediate" on at least one of the Simple 7 composite score items (e.g. not meeting Physical Activity Guidelines for Americans)
* Live in one of the designated towns in NY and TX

FFM also must:

* Provide consent electronically
* Be family members or friends identified by a CCM

CR also must:

* Provide consent electronically
* Live in one of the designated towns in NY and TX

Exclusion Criteria:

* Cognitive impairment (if it precludes completion of assessments and/or intervention)
* Inability to communicate due to severe, uncorrectable hearing loss or speech disorder (if it precludes completion of assessments and/or intervention)
* Severe visual impairment (if it precludes completion of assessments and/or intervention)
* Inability to read (as it precludes completion of assessments and/or intervention)
* Already included in another study sample (e.g. CR cannot also be CCM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2420 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in American Heart Association's Life's Simple 7 (LS7) cardiovascular health score | Baseline to 24 months
  American Heart Association's Life's Simple 7 (LS7) score is a composite of cardiovascular disease (CVD) risk factors (physical activity, eating habits, smoking status, cholesterol, glucose, body mass index (BMI), and blood pressure). Score ranges from 0 to 14. Higher scores indicate better health.

SECONDARY OUTCOMES:
Change in body mass index (BMI) | Baseline to 24 months
  Height and weight will be self-measured and BMI will be calculated.
Change in waist circumference | Baseline to 24 months
  Waist circumference (cm(in)) will be self-measured.
Percent with high/elevated blood pressure | Baseline to 24 months
  Percent with high/elevated blood pressure will be classified from self-reported measurements, diagnosis, and medication use.
Percent with high/borderline high cholesterol. | Baseline to 24 months
  Percent with high/borderline high cholesterol will be classified from self-reported measurements, diagnosis, and medication use.
Percent with diabetes/prediabetes | Baseline to 24 months
  Percent with diabetes/ prediabetes will be classified from self-reported measurements, diagnosis, and medication use.
Change in general health status | Baseline to 24 months
  General health status will be assessed using the general health question from the 36-Item Short Form Survey (SF-36). Scores range from 1 to 5. Higher scores indicate better health.
Current smoker (y/n) | Baseline to 24 months
  Whether or not a participant currently smokes will be assessed using an LS7 item.
Change in total HEI score | Baseline to 24 months
  Total Healthy Eating Index (HEI) score will be calculated from a single 24-hour recall collected via the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24). Score ranges from 0 to 100. Higher scores indicate better diet.
Change in fruit and vegetable intake | Baseline to 24 months
  Total fruit and vegetable intake (cups/day) will be measured using a LS7 item and a 24-hour recall.
Change in consumption of whole grains | Baseline to 24 months
  Whole grain consumption (servings/day) will be assessed using an LS7 item and a 24-hour recall.
Change in fiber intake | Baseline to 24 months
  Fiber intake (g/day) will be assessed using the NHANES Dietary Screener Questionnaire (DSQ) and a 24-hour recall.
Met recommendation for fish consumption (y/n) | Baseline to 24 months
  Whether or not a participant met the recommendation for fish consumption will be assessed using an LS7 item.
Change in frequency of consuming ultra-processed foods | Baseline to 24 months
  Frequency of ultra-processed foods consumption (times/month) will be assessed using a 9-item questionnaire adapted from the DSQ and the Beverage and Snack Questionnaire (BSQ2) and a 24-hour recall.
Change in red and processed meat consumption | Baseline to 24 months
  Total red and processed meat consumption (g/week) will be estimated using the DSQ and a 24-hour recall.
Change in alcohol consumption | Baseline to 24 months
  Alcohol consumption (drinks/day) will be assessed using a 2-item questionnaire adapted from the Alcohol Use Disorders Screening Test (AUDIT) and a 24-hour recall.
Change in total steps per day | Baseline to 24 months
  Total steps per day will be calculated using the average of self-reported pedometer or wearable fitness tracker readings.
Change in total physical activity | Baseline to 24 months
  Total physical activity (MET-min/wk) will be assessed using the International Physical Activity Questionnaire long form (IPAQ-long).
Change in World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) recommendation adherence score | Baseline to 24 months
  WCRF/AICR recommendation adherence score is a composite of seven items listed above: BMI, physical activity, fiber intake, fruit and vegetable consumption, processed food consumption, red meat consumption, and alcohol consumption. Scores range from 0 to 7. Higher scores indicate greater adherence to the recommendations.
Change in healthy eating motivation | Baseline to 24 months
  Healthy eating motivation will be assessed by an adapted version of the Naughton & McCarthy Healthy Eating Motivation scale (3 items). Scores range from 1 to 5. Higher scores indicate greater motivation.
Change in confidence for healthy eating | Baseline to 24 months
  Confidence for healthy eating will also be assessed by using a newly created scale (7 items) adapted from the Sallis Eating Habits Confidence Survey and the Seguin-Fowler Expanded Eating Habits Confidence Survey (7 items). Scores range from 1 to 5. Higher scores indicate greater confidence.
Change in social support for healthy eating | Baseline to 24 months
  Social support (family and friends) for healthy eating will be assessed by the Ball Social Support for Healthy Eating scale. Scores range from 1 to 5. Higher scores indicate greater social support.
Change in exercise attitudes | Baseline to 24 months
  Exercise attitudes will be assessed using selected items adapted from section 2, question 5 of the AARP Exercise Attitudes and Behaviors Survey (4 items). Scores range from 1 to 5. Higher scores indicate more positive attitudes.
Change in exercise confidence | Baseline to 24 months
  Exercise confidence will be assessed by an adapted version of the Sallis Exercise Confidence Survey (3 items). Scores range from 1 to 5. Higher scores indicate greater confidence.
Change in social support for physical activity | Baseline to 24 months
  Social support (family and friends) for physical activity will be assessed by the Ball Social Support for Physical Activity scale. Scores range from 1 to 5. Higher scores indicate greater social support.
Change in social engagement | Baseline to 24 months
  Social engagement (family and friends) will be assessed by the Lubben Social Network Scale. Scores range from 1 to 5. Higher scores indicate greater social engagement.
Change in (community) social cohesion | Baseline to 24 months
  Community social cohesion will be assessed by the social cohesion sub-scale of the Mujahid et al. Neighborhood Environment Scale (NES). Scores range from 1 to 5. Higher scores indicate greater social cohesion.
Change in individual mobilization | Baseline to 24 months
  Individual mobilization will be assessed using the human capital sub-scale of the Jakes & Shannon Mobilization Scale - Individual. Scores range from 1 to 5. Higher scores indicate greater mobilization.
Change in general civic engagement attitudes | Baseline to 24 months
  Civic engagement attitudes will be assessed by the attitudes sub-scale of the Doolittle & Faul Civic Engagement Scale. Scores range from 1 to 5. Higher scores indicate more positive civic engagement attitudes.
Change in general civic engagement behaviors | Baseline to 24 months
  Civic engagement behaviors will be assessed by the behaviors sub-scale of the Doolittle & Faul Civic Engagement Scale. Scores range from 1 to 5. Higher scores indicate more frequent civic engagement behaviors.
Change in investment in community health | Baseline to 24 months
  Investment in community health (number of priorities) will be assessed using the investment in community health sub-scale of the RWJF National Survey of Health Attitudes. Scores range from 0 to 5. Higher scores indicate higher priority placed on community health.
Change in walking environment | Baseline to 24 months
  Walking environment will be assessed by an adapted walking sub-scale of the NES (7 items). Scores range from 1 to 5. Higher scores indicate more favorable walking environments.
Change in neighborhood safety | Baseline to 24 months
  Neighborhood safety will be assessed by an adapted neighborhood safety sub-scale of the NES (3 items). Scores range from 1 to 5. Higher scores indicate greater neighborhood safety.
Change in neighborhood aesthetic | Baseline to 24 months
  Neighborhood aesthetic quality will be assessed by an adapted neighborhood aesthetic sub-scale of the NES (2 items). Scores range from 1 to 5. Higher scores indicate a more favorable neighborhood.
Change in fresh fruit and vegetable availability | Baseline to 24 months
  Fresh fruit and vegetable availability will be assessed by an adapted fresh fruit and vegetable availability sub-scale (3 items) of the Green & Glanz Perceived Nutrition Environment Measures Survey (NEMS-P). Scores range from 1 to 5. Higher scores indicate greater availability.
Change in store selection motivation | Baseline to 24 months
  Store selection motivation will be assessed by an adapted store selection motivation sub-scale from NEMS-P (3 items). Scores range from 1 to 5. Higher scores indicate greater motivation.
Change in restaurant healthy food availability | Baseline to 24 months
  Restaurant healthy food availability will be assessed by an adapted restaurant healthy food availability sub-scale from NEMS-P (2 items). Scores range from 1 to 5. Higher scores indicate greater availability of healthy food in restaurants.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A. Seguin-Fowler, PhD, Principal Investigator — Texas A&M AgriLife Research
Locations (13):
- United States (13):
  - Camden and surrounding towns, Camden, New York
  - Canastota, Canastota, New York
  - Carthage and surrounding towns, Carthage, New York
  - Hamilton and surrounding towns, Hamilton, New York
  - Rome, Rome, New York
  - Hounsfield and surrounding towns, Sackets Harbor, New York
  - Watertown, Watertown, New York
  - Center and Shelbyville, Center, Texas
  - Groveton and Woodlake, Groveton, Texas
  - Littlefield and surrounding towns, Littlefield, Texas
  - Marshall, Marshall, Texas
  - Plainview, Plainview, Texas
  - Trinity, Trinity, Texas

REFERENCES:
- [Derived] Graham ML, Eldridge GD, Demment M, Kershaw M, Christou A, Luong V, Andreyeva E, Folta SC, Hanson KL, Maddock JE, Seguin-Fowler RA. Leadership Characteristics of Extension Agents Facilitating a Healthy Communities, Civic-Engagement Randomized Trial in Rural Towns. J Healthy Eat Act Living. 2024 Dec 1;4(3):174-188. eCollection 2024. PMID 40385265
- [Derived] Seguin-Fowler RA, Hanson KL, Villarreal D, Rethorst CD, Ayine P, Folta SC, Maddock JE, Patterson MS, Marshall GA, Volpe LC, Eldridge GD, Kershaw M, Luong V, Wang H, Kenkel D. Evaluation of a civic engagement approach to catalyze built environment change and promote healthy eating and physical activity among rural residents: a cluster (community) randomized controlled trial. BMC Public Health. 2022 Sep 4;22(1):1674. doi: 10.1186/s12889-022-13653-4. PMID 36058913